CLINICAL TRIAL: NCT01643031
Title: Effect of Modifying Anti-platelet Treatment to Ticagrelor in Patients With Diabetes and Low Response to Clopidogrel
Acronym: MATTIS-D
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Tel Aviv Medical Center (Other); Sheba Medical Center (Other Government); Meir Medical Center (Other); Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, eli lev, Prof. Eli Lev, Director, Cardiac catheterization laboratory, Hasharon Hospital, Rabin Medical Center, Israel, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6793
Record Dates: First submitted 2012-07-15; First posted 2012-07-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes Mellitus; Coronary Disease
Keywords: Diabetes; Platelets aggregation inhibitors; Platelet function tests
MeSH Terms: conditions — Diabetes Mellitus; Coronary Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental): Patients randomized to the ticagrelor group will receive ticagrelor at a dose of 180 mg given 1-2 hours before the coronary angiography, followed by 90 mg twice a day for 30 days after the PCI. After 30 days the patient will be invited to a special research clinic in the hospital and his treatment will be switched back to clopidogrel (to complete 1 year of treatment).
  Interventions: Drug: Ticagrelor
- Continued Clopidogrel (Active Comparator): Patients randomized to continued clopidogrel treatment will be given an additional 300 mg of clopidogrel loading 1-2 hours before coronary angiography (in addition to the previous 300 mg load or chronic clopidogrel therapy the patient received), followed by 75 mg a day for 1 year after the PCI
  Interventions: Drug: Continued clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor will be given (to patients with low response to clopidogrel randomized to the Ticagrelor group) at a dose of 180 mg given 1-2 hours before the coronary angiography, followed by 90 mg twice a day for 30 days after the PCI. After 30 days the patient's treatment will be switched back to clopidogrel (to complete 1 year of treatment).
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Continued clopidogrel — Patients with low response to clopidogrel randomized to continued clopidogrel treatment will be given an additional 300 mg of clopidogrel loading 1-2 hours before coronary angiography (in addition to the previous 300 mg load or chronic clopidogrel therapy the patient received), followed by 75 mg a day for 1 year after the PCI
  Other Names: Plavix
  Arms: Continued Clopidogrel

SUMMARY:
In recent years numerous studies have shown that the response of patients to the anti-platelet drug clopidogrel is widely variable. Furthermore, patients who do not respond well to the drug ("resistant") have been shown to be at increased risk to develop cardiac events, including myocardial infarction and mortality. It thus seems reasonable to test the efficacy of the drug (by platelet function tests) and modify treatment accordingly. However, a large study that examined a strategy of routine testing of clopidogrel response in thousands of patients (GRAVITAS study) did not show any clinical benefit. This study was limited, however, by a very low event rate (2.3%), and by the strategy employed to treat patients with low response (increasing the clopidogrel dose), which is currently known to be ineffective in many patients with low response. To overcome these limitations the investigators plan to examine a high risk population - patients with diabetes planned to undergo coronary angiography - and to treat clopidogrel low responders by switching their treatment to the potent anti-platelet drug ticagrelor, which has been shown to overcome clopidogrel low response.

The investigators hypothesize that patients with diabetes and low response to clopidogrel will benefit clinically from switching therapy to ticagrelor. The main endpoint of the study will be the risk of myocardial enzyme elevation following percutaneous coronary intervention (PCI); a marker which has been strongly associated with poor clinical outcome.

The aim of the study is, therefore, to assess whether a strategy of monitoring platelet function during clopidogrel treatment in patients with diabetes undergoing PCI, and modifying treatment to ticagrelor in patients with low response, will be associated with reduced risk of myocardial enzyme release.

The investigators plan to enroll patients with treated diabetes, planned to undergo coronary angiography. Patients with acute or recent myocardial infarction will be excluded. They will be tested for response to clopidogrel by the VerifyNow P2Y12 assay (either on chronic clopidogrel treatment or 12-24 hours after receiving 300 mg clopidogrel). Patients with low response to clopidogrel (≥ 208 PRU) will be randomized to either continued treatment with clopidogrel (75 mg/day), or switching of treatment to ticagrelor (90 mg twice a day) for 30 days (followed by continued clopidogrel therapy). The primary endpoint will be the rate of troponin of CK-MB (cardiac enzymes) measured 20-24 hours after the PCI. Secondary endpoints will be the occurrence of adverse clinical endpoints - myocardial infarction, need for urgent revascularization or mortality at 30 days. The investigators aim to enroll 100 patients in each study group (ticagrelor vs. continued clopidogrel). Assuming a clopidogrel low response rate of 40% among patients with diabetes, about 500 patients would have to be screened to identify 200 patients with low response.

DETAILED DESCRIPTION:
BACKGOUND The concept of monitoring platelet reactivity in patients treated with clopidogrel and tailoring treatment according to the results has been under intense debate in recent years. There is clear and consistent evidence that there is wide variability in the anti-platelet response to clopidogrel, and that patients with low response (more accurately termed - high on treatment platelet reactivity) are at increased risk of adverse cardiac events - mainly stent thrombosis and myocardial infarction. However, the only large randomized trial that examined a strategy of routing monitoring of platelet reactivity and response to clopidogrel and tailoring treatment accordingly (by increasing the clopidogrel maintenance dose) - the GRAVITAS study - was negative. Thus, although from a physiological perspective it seems reasonable to monitor the effects of a drug with such wide variability (and poor prognosis associated with low response), clinical evidence in support of routine monitoring is lacking. When analyzing the negative results of the GRAVITAS study, two main factors should be discussed: a very low clinical adverse event rate (2.3% in each of study the groups) probably reflecting a low risk patient population, and the strategy chosen to overcome high on treatment platelet reactivity (HTPR) - increasing the maintenance clopidogrel dose from 75 mg daily to 150 mg daily, which is currently known to be ineffective in overcoming clopidogrel HTPR in many of the patients.

In light of these potential limitations of the GRAVITAS study the investigators propose a study based on the following aspects:

1. A potent strategy to overcome clopidogrel HTPR - treatment with ticagrelor, which has been clearly shown to overcome low response to clopidogrel.
2. Higher risk population - only patients with treated diabetes (shown in the BARI-2D study to have a 10-12% rate of major cardiovascular events at 1 year).
3. Rather than a composite clinical endpoint, the primary endpoint will be the rate of CK-MB or troponin elevation following percutaneous coronary intervention (PCI), which has been consistently associated with a higher risk of cardiovascular adverse events, and occurs at a rate of about 35% in patients with low response to clopidogrel.

The aim of the study is to assess whether a strategy of monitoring platelet reactivity during clopidogrel treatment in patients with diabetes undergoing PCI, and modifying the treatment to ticagrelor in patients with HTPR, is associated with a lower rate of myocardial enzyme elevation following PCI.

METHODS

See inclusion and exclusion criteria in the following sections.

Patients treated chronically with clopidogrel 75 mg per day will undergo platelet function testing under this treatment regimen. Patients who are clopidogrel naïve will be given 300 mg loading of clopidogrel and be tested about 12-24 hours after this loading dose. For all patients, platelet function testing will be performed before the coronary angiography.

Platelet function testing will be performed with the VerifyNow P2Y12 assay (Accumetrics Inc.), using a cutoff value of ≥ 208 reaction units to define HTPR.

Patients with HTPR will be randomized 1:1 to receive either ticagrelor or additional clopidogrel.

Ticagrelor regimen: 180 mg given 1-2 hours before the coronary angiography, followed by 90 mg twice a day for 30 days in case PCI was performed. After 30 days the patient will be invited to a special research clinic in the hospital and his treatment will be switched to clopidogrel (with 300 mg loading, and 75 mg a day thereafter for 11 additional months - for a total period of 1 year). The 30 day ticagrelor period was chosen because prior studies have shown that platelet hyper-reactivity and low response to clopidogrel are prominent in the first days after PCI, and subside significantly within 30 days after the procedure. In addition, most cases of stent thrombosis occur in the first month following PCI.

Clopidogrel regimen: 300 mg given 1-2 hours before coronary angiography (in addition to the previous 300 mg load or chronic clopidogrel therapy the patient received), followed by 75 mg a day for 1 year case PCI was performed.

The investigators aim to enroll a total of 200 patients with HTPR who will undergo PCI - 100 patients in each group (ticagrelor vs. continued clopidogrel). Patients who will not undergo PCI will be withdrawn from the study.

Choice of stent during PCI will be left to the operator's discretion, but given the diabetes status of all patients, use of drug eluting stents will be encouraged. PCI will be performed according to standard practice and operator preferences (regarding to access, pre- and post dilatation etc.). Use of glycoprotein IIb/IIIa inhibitors will be discouraged, unless in bailout situations. Patients who will receive glycoprotein IIb/IIIa inhibitors will be excluded from the analysis.

An additional VerifyNow P2Y12 test will be performed in the 200 patients with initial HTPR, 20-24 hours following the PCI; at this time point troponin and CK-MB levels will also be evaluated.

Primary endpoint: rate of elevation of troponin or CK-MB (above the upper limit of normal, and above 3 times the upper limit of normal) measured 20-24 hours after the PCI.

Secondary endpoint: rate of major adverse cardiovascular endpoints including death, myocardial infarction or urgent target vessel revascularization at 30 days.

Sample size calculation: assuming a rate of CK-MB or troponin elevation post-PCI of 35% among patients with low response to clopidogrel, 100 patients in each group would allow detection of a 50% difference in the primary endpoint between the groups (50% reduction in myocardial enzyme elevation rate with ticagrelor), with an alpha of 0.05 and power of 0.80. Assuming a HTPR rate of 40% using the 208 VerifyNow cutoff value, 500 patients would have to be screened in order to identify 200 patients with HTPR (not taking into consideration the patients that would not require PCI and be withdrawn from the study).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diabetes treated with oral hypoglycemic medications and/or insulin.
2. Aged 30-80 years.
3. Patients with stable angina and a positive non-invasive test, or patients with unstable angina, all planned to undergo coronary angiography.
4. Treated with aspirin 75-100 mg per day.

   -

Exclusion Criteria:

1. Any myocardial infarction (STEMI or non-STEMI) as the indication for the cardiac catheterization. Thus, only troponin-negative and CK-MB negative patients will be included.
2. Any contraindications to ticagrelor or clopidogrel.
3. Anemia (Hg<10 g/dL) or thrombocytopenia (<100,000 / mm3)
4. Chronic renal failure (Cr ≥ 2.5 mg/dL)

   -

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Rate of elevation of troponin or CK-MB (above the upper limit of normal, and above 3 times the upper limit of normal) measured 20-24 hours after the PCI. | 20-24 hours after the PCI
  Rate of elevation of troponin or CK-MB (above the upper limit of normal, and above 3 times the upper limit of normal) measured 20-24 hours after the PCI.

SECONDARY OUTCOMES:
Rate of major adverse cardiovascular endpoints including death, myocardial infarction or urgent target vessel revascularization at 30 days | 30 days
  Rate of major adverse cardiovascular endpoints including death, myocardial infarction or urgent target vessel revascularization at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Eli I Lev, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Bonello L, Tantry US, Marcucci R, Blindt R, Angiolillo DJ, Becker R, Bhatt DL, Cattaneo M, Collet JP, Cuisset T, Gachet C, Montalescot G, Jennings LK, Kereiakes D, Sibbing D, Trenk D, Van Werkum JW, Paganelli F, Price MJ, Waksman R, Gurbel PA; Working Group on High On-Treatment Platelet Reactivity. Consensus and future directions on the definition of high on-treatment platelet reactivity to adenosine diphosphate. J Am Coll Cardiol. 2010 Sep 14;56(12):919-33. doi: 10.1016/j.jacc.2010.04.047. PMID 20828644
- [Background] Price MJ, Berger PB, Teirstein PS, Tanguay JF, Angiolillo DJ, Spriggs D, Puri S, Robbins M, Garratt KN, Bertrand OF, Stillabower ME, Aragon JR, Kandzari DE, Stinis CT, Lee MS, Manoukian SV, Cannon CP, Schork NJ, Topol EJ; GRAVITAS Investigators. Standard- vs high-dose clopidogrel based on platelet function testing after percutaneous coronary intervention: the GRAVITAS randomized trial. JAMA. 2011 Mar 16;305(11):1097-105. doi: 10.1001/jama.2011.290. PMID 21406646
- [Background] Oestreich JH, Holt J, Dunn SP, Smyth SS, Campbell CL, Charnigo R, Akers WS, Steinhubl SR. Considerable variability in platelet activity among patients with coronary artery disease in response to an increased maintenance dose of clopidogrel. Coron Artery Dis. 2009 May;20(3):207-13. doi: 10.1097/MCA.0b013e328329924b. PMID 19318928
- [Background] Gladding P, Webster M, Zeng I, Farrell H, Stewart J, Ruygrok P, Ormiston J, El-Jack S, Armstrong G, Kay P, Scott D, Gunes A, Dahl ML. The antiplatelet effect of higher loading and maintenance dose regimens of clopidogrel: the PRINC (Plavix Response in Coronary Intervention) trial. JACC Cardiovasc Interv. 2008 Dec;1(6):612-9. doi: 10.1016/j.jcin.2008.09.005. PMID 19463374
- [Background] Gurbel PA, Bliden KP, Butler K, Antonino MJ, Wei C, Teng R, Rasmussen L, Storey RF, Nielsen T, Eikelboom JW, Sabe-Affaki G, Husted S, Kereiakes DJ, Henderson D, Patel DV, Tantry US. Response to ticagrelor in clopidogrel nonresponders and responders and effect of switching therapies: the RESPOND study. Circulation. 2010 Mar 16;121(10):1188-99. doi: 10.1161/CIRCULATIONAHA.109.919456. Epub 2010 Mar 1. PMID 20194878
- [Background] BARI 2D Study Group; Frye RL, August P, Brooks MM, Hardison RM, Kelsey SF, MacGregor JM, Orchard TJ, Chaitman BR, Genuth SM, Goldberg SH, Hlatky MA, Jones TL, Molitch ME, Nesto RW, Sako EY, Sobel BE. A randomized trial of therapies for type 2 diabetes and coronary artery disease. N Engl J Med. 2009 Jun 11;360(24):2503-15. doi: 10.1056/NEJMoa0805796. Epub 2009 Jun 7. PMID 19502645
- [Background] Feldman DN, Kim L, Rene AG, Minutello RM, Bergman G, Wong SC. Prognostic value of cardiac troponin-I or troponin-T elevation following nonemergent percutaneous coronary intervention: a meta-analysis. Catheter Cardiovasc Interv. 2011 Jun 1;77(7):1020-30. doi: 10.1002/ccd.22962. Epub 2011 May 13. PMID 21574239
- [Background] Nienhuis MB, Ottervanger JP, Bilo HJ, Dikkeschei BD, Zijlstra F. Prognostic value of troponin after elective percutaneous coronary intervention: A meta-analysis. Catheter Cardiovasc Interv. 2008 Feb 15;71(3):318-24. doi: 10.1002/ccd.21345. PMID 18288753
- [Background] Lev EI, Patel RT, Maresh KJ, Guthikonda S, Granada J, DeLao T, Bray PF, Kleiman NS. Aspirin and clopidogrel drug response in patients undergoing percutaneous coronary intervention: the role of dual drug resistance. J Am Coll Cardiol. 2006 Jan 3;47(1):27-33. doi: 10.1016/j.jacc.2005.08.058. Epub 2005 Dec 9. PMID 16386660
- [Background] Price MJ, Angiolillo DJ, Teirstein PS, Lillie E, Manoukian SV, Berger PB, Tanguay JF, Cannon CP, Topol EJ. Platelet reactivity and cardiovascular outcomes after percutaneous coronary intervention: a time-dependent analysis of the Gauging Responsiveness with a VerifyNow P2Y12 assay: Impact on Thrombosis and Safety (GRAVITAS) trial. Circulation. 2011 Sep 6;124(10):1132-7. doi: 10.1161/CIRCULATIONAHA.111.029165. Epub 2011 Aug 29. PMID 21875913
- [Background] Campo G, Parrinello G, Ferraresi P, Lunghi B, Tebaldi M, Miccoli M, Marchesini J, Bernardi F, Ferrari R, Valgimigli M. Prospective evaluation of on-clopidogrel platelet reactivity over time in patients treated with percutaneous coronary intervention relationship with gene polymorphisms and clinical outcome. J Am Coll Cardiol. 2011 Jun 21;57(25):2474-83. doi: 10.1016/j.jacc.2010.12.047. PMID 21679849
- [Background] Gurbel PA, Bliden KP, Hiatt BL, O'Connor CM. Clopidogrel for coronary stenting: response variability, drug resistance, and the effect of pretreatment platelet reactivity. Circulation. 2003 Jun 17;107(23):2908-13. doi: 10.1161/01.CIR.0000072771.11429.83. Epub 2003 Jun 9. PMID 12796140